CLINICAL TRIAL: NCT04479033
Title: Caring for Persons With Dementia and Their Caregivers in the Community: Towards a Sustainable Community Based Dementia Care System
Brief Title: Caring for Persons With Dementia and Their Caregivers in the Community
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Ministry of Health, Singapore (Other Government); The Tsao Foundation (Unknown)
Responsible Party: Principal Investigator, Angelique Chan, Executive Director, Duke-NUS Graduate Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOH/NIC/COG05/2017-00
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Dementia; Cognitive Impairment
Keywords: community based care; multidisciplinary team; comprehensive needs assessment; moderate to severe dementia; mixed-methods evaluation
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants assigned to the control group had screened positive for cognitive impairment but refused the intervention. They were provided with a GP referral letter and information on helplines and caregiver support. Follow-up interviews were scheduled at week 24.
- Intervention (Experimental): Weekly meeting/communication sessions with members of intervention team for a total of 24 weeks.
  Interventions: Other: Multidisciplinary collaborative model of community care management

INTERVENTIONS:
Other: Multidisciplinary collaborative model of community care management — An individualised care plan is developed for PLWDs-caregiver dyads who meet/communicate weekly with various members of the HMDCS team depending on the nature of their needs. Each dyad's care plan involves the diagnosis of problems (eg: memory problems, family conflicts, poor nutrition, fall risk, medication compliance, lack of long-term care arrangements), establishment of treatment goals (eg: caregiver education, awareness of long-term care planning, stabilising medical care at home, improving emotional support), and indicating specific interventions (eg: referrals to counsellors, specialist doctors, day rehabilitation centres; consultations at GP clinic; coordination of advanced care planning; installation of home safety devices; training caregivers to detect acute deterioration in PLWDs). Monitoring of the dyads' statuses and updating of care plans are performed throughout the duration of the programme.
  Arms: Intervention

SUMMARY:
The study consists of two phases - i) a comprehensive assessment of biopsychosocial needs among cognitively impaired persons and their family caregivers residing in the Whampoa residential estate in Singapore ; ii) a quasi-experimental evaluation of a pilot community-based dementia care programme administered by a multidisciplinary team of service providers. The intervention is a physician-enhanced dementia-specific care management programme that supports client dyads for up to six months and through community care management, person-centred communication, management of challenging behaviours, psychoeducation, geriatric medicine, and gerontological approaches. The intervention team consists of a nurse, social worker, care manager, physician, and 'Dementia Care Program Assistants' who specifically design personalised meaningful activities to engage persons living with dementia as well as provide caregivers with training in basic dementia caregiving.

DETAILED DESCRIPTION:
To provide appropriate care for persons living with dementia (PLWDs) in the community, their needs (met, unmet, and latent) and that of their caregivers must be understood holistically. Local studies have yet to comprehensively examine the experiences of community dwelling older persons living with moderate to severe dementia and their caregivers, and the impact of an integrated community model of health care and psychosocial support. This study adopts a mixed-method approach to needs assessment and programme evaluation using qualitative in-depth interviews and quantitative surveys administered to participants assigned to control and intervention groups. The Hua-Mei Dementia Care System (HMDCS) is a programme that aims to empower and support both PLWDs and their caregivers through personalised care management, dementia-specific education, and cognitive training. The HMDCS addresses the multifaceted challenges faced by PLWD-caregiver dyads such as behavioural problems, psychological distress, lack of social participation, stigma, communication barriers, financial strain, and insufficient social support.

The study aims are to:

1. Explore the perceptions, behaviours, and underlying motivators and inhibitors of PLWDs, their caregivers, and members of the community
2. Assess the health, social, psychological, and emotional needs of community dwelling PLWDs and their caregivers
3. Evaluate the effectiveness of the programme in reducing cognitive and functional decline, caregiver burden, as well as improving self-reported health status, social wellbeing, and quality of life of PLWD-caregiver dyads

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age and above.
* Singapore citizens or permanent residents.
* Lives within catchment area of Whampoa Constituency
* Screened positively for cognitive impairment (MMSE score of 15 and above)
* PLWDs must have a primary caregiver.
* Caregivers must be 21 years of age and above.

Exclusion Criteria:

• PLWDs without a caregiver

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-04-27 (Actual); Primary Completion 2021-02-27 (Estimated); Study Completion 2021-02-27 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in cognitive impairment at week 24. | Baseline, Week 24
  Mini-Mental State Examination is a 30-point test to screen for cognitive impairment. Scores ranging from 20 to 26 indicate some cognitive impairment, 10-19 indicate moderate to severe cognitive impairment and below 10 indicate very severe cognitive impairment.
Change from baseline in caregiver stress and burden at week 24. | Baseline, Week 24
  Zarit Burden Interview is a 22-item instrument for measuring the caregiver's perceived burden of providing care. Questions focus on caregiver's health, psychological well-being, finances, social life and relationship between the caregiver and the PLWD.
Change from baseline in memory and behaviour problems at week 24. | Baseline, Week 24
  Revised Memory and Behavior Problems Checklist is a 24-item (scored on a scale of 0-4) caregiver-report to measure behavioral problems in PLWDs. The items can be summed as a total score and 3 subscale scores in the domains of memory, depression, and disruptive behaviors. Parallel scores for caregiver reaction are also obtained. Such disruptive and challenging behaviors undermine quality of life in PWDs and place both an emotional and financial burden on their caregivers.
Change from baseline in health-related quality of life at week 24. | Baseline, Week 24
  Euro-Qol-5D- EQ5D is a commonly used 5-item scale to measure health-related quality of life.

SECONDARY OUTCOMES:
Cost-effectiveness of intervention | Baseline, Week 24
  Cost-effectiveness of the new model of care will be assessed using the incremental cost-effectiveness ratio (ICER) with respect to the control group. Cost will be assessed by recording utilization of health care and long-term care services and their average unit costs. The calculated ICER will show the cost of a quality-adjusted life year (QALY) saved by the new model of care. Effectiveness will be assessed by computing the average quality-adjusted life years left to live by the dementia participant in both groups. As the intervention is not assumed to be life-extending, study groups will only differ through their quality of life as measured by EQ5D weights. We will account for the quality of life of both PLWDs and their caregivers and sum their respective contributions.

CONTACTS AND LOCATIONS:
Overall Officials: Angelique Chan, PhD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Medical School, Singapore, Singapore